CLINICAL TRIAL: NCT01896349
Title: Efficacy of Interpersonal Psychotherapy in Treatment Resistant Depression
Brief Title: Interpersonal Psychotherapy for Treatment Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIP-120288
Record Dates: First submitted 2013-07-01; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Treatment Resistant Depression
Keywords: Psychotherapy, Treatment Resistant Depression, depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Interpersonal Psychotherapy; Antidepressive Agents; Fluoxetine; Sertraline; Paroxetine; Citalopram; Escitalopram; Fluvoxamine; Venlafaxine Hydrochloride; Duloxetine Hydrochloride; Bupropion; Lithium; Risperidone; Tranylcypromine; Imipramine; Amitriptyline; Clomipramine; Nortriptyline; Trazodone; Mirtazapine; Sulpiride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPT+antidepressant drugs (Experimental): Interpersonal Psychotherapy protocol (IPT) consist of 16 sessions of manualized interpersonal psychotherapy for depression. Patients are allowed to reschedule 3 sessions if they miss their appointments.
  Antidepressant Drugs protocol consist of pharmacological management of depression, oriented by international guidelines, clinician´s free choice. Monotherapy or combinations are allowed. Antidepressant and drugs are: fluoxetine, sertraline, paroxetin, citalopram, escitalopram, fluvoxamine, venlafaxin, duloxetin, bupropion, lithium, risperidone, tranylcypromine, Imipramine, amitriptyline, clomipramine, nortriptyline, trazodone, mirtazapine, sulpiride.
  Interventions: Other: IPT+ antidepressant drugs; Drug: fluoxetine; Drug: sertraline; Drug: paroxetine; Drug: Citalopram; Drug: escitalopram; Drug: fluvoxamine; Drug: Venlafaxine; Drug: Duloxetine; Drug: Bupropion; Drug: Lithium; Drug: Risperidone; Drug: tranylcypromine; Drug: Imipramine; Drug: amitriptyline; Drug: Clomipramine; Drug: nortriptyline; Drug: trazodone; Drug: Mirtazapine; Drug: sulpiride
- Antidepressant Drugs (Active Comparator): Drugs protocol consist of pharmacological management of depression, oriented by international guidelines, clinician´s free choice.
  Antidepressant Drugs protocol consist of pharmacological management of depression, oriented by international guidelines, clinician´s free choice. Monotherapy or combinations are allowed. Antidepressant and drugs are: fluoxetine, sertraline, paroxetine, citalopram, escitalopram, fluvoxamine, venlafaxine, duloxetine, bupropion, lithium, risperidone, tranylcypromine, Imipramine, amitriptyline, clomipramine, nortriptyline, trazodone, mirtazapine, sulpiride.
  Interventions: Drug: fluoxetine; Drug: sertraline; Drug: paroxetine; Drug: Citalopram; Drug: escitalopram; Drug: fluvoxamine; Drug: Venlafaxine; Drug: Duloxetine; Drug: Bupropion; Drug: Lithium; Drug: Risperidone; Drug: tranylcypromine; Drug: Imipramine; Drug: amitriptyline; Drug: Clomipramine; Drug: nortriptyline; Drug: trazodone; Drug: Mirtazapine; Drug: sulpiride

INTERVENTIONS:
Other: IPT+ antidepressant drugs — 16 sessions of interpersonal psychotherapy plus antidepressant drugs.
  Other Names: Interpersonal Psychotherapy; Antidepressant drugs
  Arms: IPT+antidepressant drugs
Drug: fluoxetine — Antidepressant drugs, clinician´s free choice oriented by guidelines. Monotherapy or combinations are allowed
Drug: sertraline
Drug: paroxetine
Drug: Citalopram
Drug: escitalopram
Drug: fluvoxamine
Drug: Venlafaxine
Drug: Duloxetine
Drug: Bupropion
Drug: Lithium
Drug: Risperidone
Drug: tranylcypromine
Drug: Imipramine
Drug: amitriptyline
Drug: Clomipramine
Drug: nortriptyline
Drug: trazodone
Drug: Mirtazapine
Drug: sulpiride

SUMMARY:
The purpose of this study is to determine whether combination of antidepressant drugs plus interpersonal psychotherapy is superior to antidepressant drugs alone in treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnose of unipolar treatment resistant depression

Exclusion Criteria:

* Patients diagnose of: bipolar disorder, psychosis, high suicide risk, Intellectual disability, illicit drug dependence.
* Currently in or having received psychotherapy in the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-08 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) - continuous | End point week 19 and Week 24
  Score change on Hamilton depression scale from baseline to week 19 and to week 24

SECONDARY OUTCOMES:
Beck depression Inventory (BDI) | End point week 19 and Week 24
  Score change on Beck depression inventory from baseline to week 19 and to week 24

OTHER OUTCOMES:
Clinical Global Impression - Severity Scale (CGI-S) / dichotomous | Endpoint (week-19) and week 24
Whoqol brief - World Health Organization Quality of Life Instrument - Short version - Brazilian version | Endpoint week 19 and week 24
  Score change in Whoqol-breef from baseline to week 19 and week 24
Biological measures - BDFN, TBARS, TNF-alfa, IL-1, IL-6 | End point week 19 and Week 24
  A blood sample will be collected at baseline, week 19 and week 24. Change in serum biomarkers will be evaluated - BDFN (Brain derived neurotrophic factor), TBARS (thiobarbituric acid reactive substance), TNF-alfa (tumor necrosis factor alfa), IL-1 (interleukin-1), IL-6 (interlekin-6) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo PA Fleck, MD,PhD, Principal Investigator — Federal University of Rio Grande do Sul / Hospital de Clínicas de Porto Alegre
Locations (1):
- Federal University of Rio Grande do Sul / Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Souza LH, Salum GA, Mosqueiro BP, Caldieraro MA, Guerra TA, Fleck MP. Interpersonal psychotherapy as add-on for treatment-resistant depression: A pragmatic randomized controlled trial. J Affect Disord. 2016 Mar 15;193:373-80. doi: 10.1016/j.jad.2016.01.004. Epub 2016 Jan 8. PMID 26799332